CLINICAL TRIAL: NCT00000239
Title: Buprenorphine Pharmacology Related to Addiction Treatment
Brief Title: Buprenorphine Pharmacology Related to Addiction Treatment - 21
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: University of Vermont (Other)
Purpose: Treatment
Other Study IDs: NIDA-06969-21; R01-06969-21
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2005-08-17 (Estimated); Status verified 2002-12

CONDITIONS: Opioid-Related Disorders
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine

INTERVENTIONS:
Drug: Buprenorphine

SUMMARY:
The purpose of this study is to examine if chronic buprenorphine administration will generate supersensitivity to opiates.

ELIGIBILITY:
Please contact site for information.

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0

PRIMARY OUTCOMES:
Drug use
Opioid agonist effects
Opiate withdrawal
Physiological changes in: pupil diameter, blood pressure, heart rate, respiration

CONTACTS AND LOCATIONS:
Overall Officials: Warren Bickel, Ph.D., Principal Investigator — University of Vermont
Locations (1):
- Treatment Research Center, Burlington, Vermont, United States

REFERENCES:
- [Background] Bickel, Amass (1995 Experimental & Clinical Psychopharmacology. 3: 477-489 Amass et al 91996) Journal of Substance Abuse Treatment. 13: 43-49 Madden et al., (1997) Experimental & Clinical Psychopharmacology. 5: 1-7. Bickel, Amass (1995) Experimental & Clinical Psychopharmacology. 3: 477-489. Amass et al., (1996) Journal of Substance Abuse Treatment. 13:43-49. Madden et al., (1997) ) Experimental & Clinical Psychopharmacology. 5:1-7.